CLINICAL TRIAL: NCT02809287
Title: A Novel Laparoscopic Hepatectomy Posture, Left Lateral Position Plus Jackknife
Brief Title: A Novel Laparoscopic Hepatectomy Posture, Left Lateral Position Plus Jackknife Position
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongguo Zhou, Dr, Sun Yat-sen University
Other Study IDs: 20160609
Record Dates: First submitted 2016-06-16; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- study group: patients with left lateral position plus jackknife posture when perform laparoscopic hepatectomy
  Interventions: Procedure: Jackknife posture

INTERVENTIONS:
Procedure: Jackknife posture — patients with left lateral position plus jackknife position when perform laparoscopic hepatectomy

SUMMARY:
Since the first report of laparoscopic resection of a benign hepatic tumor by Professor H. Reith in 1991, the laparoscope has been widely used in liver disease. Based on its advantages in laparoscopic vision and amplification, laparoscopic hepatectomy (LH) has been well recognized globally. Generally speaking, for lesions located in the left, front or lower part of the liver, corresponding to Couinaud segments II, III, IVb, V and VI, an LH surgery is recommended; however, for lesions located in segments VII and VIII, the surgery is high technically difficult due to poor exposure. Therefore,the investigators employ the left lateral position plus jackknife position to better expose lesions in these segments, hoping to reduce surgical time and bleeding in LH.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were diagnosed with hepatocellular carcinoma (HCC) based on the criteria established by the European Association for the Study of the Liver
2. Tumor located in segment VI, VII, or VIII.

Exclusion Criteria:

1. Major vessel or bile duct tumor invasion,
2. Recurrent HCC
3. Tumor close to secondary vessels and bile ducts
4. Patients with extrahepatic metastasis
5. Grade C liver function,
6. Significant surgical contraindications

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were diagnosed with hepatocellular carcinoma (HCC) based on the criteria established by the European Association for the Study of the Liver
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Operation time | intraoperative
  evaluate the efficiency with this posture
Blood loss | intraoperative
  evaluate the blood loss with this posture

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen JC, Zhang RX, Chen MS, Xu L, Chen JB, Yang KL, Zhang YJ, Zhou ZG. Left jackknife position: a novel position for laparoscopic hepatectomy. Chin J Cancer. 2017 Mar 20;36(1):31. doi: 10.1186/s40880-017-0190-y. PMID 28320486